CLINICAL TRIAL: NCT03878823
Title: Safety and Pharmacokinetics of ODM-209 in Patients With Metastatic Castration-resistant Prostate Cancer or Estrogen Receptor-positive, Human Epidermal Growth Factor Receptor 2-negative Advanced Breast Cancer
Brief Title: Safety and Pharmacokinetics of ODM-209
Acronym: STESIDES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3125001
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer Metastatic; Advanced Breast Cancer; Castration-resistant Prostate Cancer; Metastatic Breast Cancer
Keywords: metastatic castration-resistant prostate cancer; advanced hormone receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ODM-209 Part 1 Dose escalation (Experimental)
  Interventions: Drug: ODM-209
- ODM-209 Part 2 Dose expansion (Experimental)
  Interventions: Drug: ODM-209

INTERVENTIONS:
Drug: ODM-209 — co-administered with glucocorticoid and mineralocorticoid, orally daily

SUMMARY:
The purpose of this first-in-human study is to evaluate safety and tolerability of ODM-209 and find the dose of ODM-209.

DETAILED DESCRIPTION:
Part 1: to evaluate the safety and tolerability of ODM-209, to define the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of ODM-209, if feasible, to define the recommended dose of ODM-209 and replacement therapy for Part 2 of the study.

Part 2: to further evaluate the safety and tolerability of ODM-209, to evaluate the preliminary anticancer activity of ODM-209.

ELIGIBILITY:
MAIN INCLUSION CRITERIA:

* Written informed consent (IC) obtained.
* Age ≥ 18 years.
* ECOG performance status 0-1.
* Adequate marrow, liver and kidney function.
* Able to swallow study treatment.

Main Prostate cancer specific inclusion criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Castration resistant prostate cancer with serum testosterone < 50 ng/dl.
* Metastatic disease.
* Ongoing androgen deprivation therapy with GnRH analogue, or have had bilateral orchiectomy.
* Have had treatment with at least one line of second generation androgen receptor targeting therapy and one line of chemotherapy.

Main Breast cancer specific inclusion criteria:

* Histologically confirmed breast carcinoma
* ER positive, HER2-negative advanced breast cancer
* Postmenopausal or pre/perimenopausal if amendable to be treated with GnRH agonist or antagonist.
* Documented disease progression after treatment with at least 2 lines of systemic treatment for advanced breast cancer. Of these, at least one line must have been endocrine treatment in combination with a cdk4/6 inhibitor.

MAIN EXCLUSION CRITERIA

* History of pituitary dysfunction.
* Known brain metastases or active leptomeningeal disease.
* Active infection or other medical condition that would make corticosteroids contraindicated.
* Hypotension or uncontrolled hypertension.
* Clinically significant cardiovascular disease, e.g. myocardial infarction, arterial thrombotic events, or pulmonary embolism in the past six months, unstable angina, or congestive heart failure (New York Heart Association [NYHA] class II-IV).
* Prolonged QTcF interval.
* Use of any investigational drug 4 weeks prior to the start of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Within first 28 days of treatment
  Highest dose level at which under 33% of patients in a cohort experience DLT

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Hänninen, Study Director — Orion Corporation, Orion Pharma
Locations (4):
- Rigshospitalet, University Hospital of Copenhagen, Copenhagen, Denmark
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Institut Gustave Roussy, Villejuif, France